CLINICAL TRIAL: NCT06344806
Title: The Effect of Breastfeeding Education Through Gamification on Breastfeeding Self-Efficacy and Infant Nutrition Attitudes of Pregnant Women: A Randomized Controlled Study
Brief Title: The Effect of Gamification on Breastfeeding Self-Efficacy and Infant Nutrition Attitudes of Pregnant Women
Acronym: gamification
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lokman Hekim University (Other Government)
Responsible Party: Principal Investigator, Özlem Ülkü BULUT, Lecturer PhD, Lokman Hekim University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: oyunlastirmabeslenme
Record Dates: First submitted 2024-03-22; First posted 2024-04-03 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Breastfeeding
Keywords: breastfeeding; gamification; education
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Gamified Breastfeeding Education (Experimental): Participants in this arm receive a structured breastfeeding education program delivered through a digital platform incorporating gamification elements during the last trimester of pregnancy.
  Interventions: Behavioral: Gamified Breastfeeding Education
- Standard Antenatal Breastfeeding Education (Active Comparator): Participants in this arm receive routine breastfeeding education provided as part of standard antenatal care services at the hospital.
  Interventions: Behavioral: Gamified Breastfeeding Education

INTERVENTIONS:
Behavioral: Gamified Breastfeeding Education — Breastfeeding education content will be integrated into the game program designed with the gamification technique. A training program will be applied to the women in the experimental group in the last trimester. Women in the control group will receive the standard breastfeeding training in the hospital. Measurement tools will be applied to all participants before and after the training.

SUMMARY:
This study aimed to evaluate the effect of a gamification-based breastfeeding education program on breastfeeding self-efficacy and infant feeding attitudes among pregnant women. The study was designed as a randomized controlled, pretest-posttest, parallel-group trial and was conducted in the antenatal outpatient clinics of Lokman Hekim Etlik Hospital.

Eligible pregnant women were randomly assigned to either an intervention group or a control group. The intervention group received breastfeeding education delivered through a digital gamification-based program during the last trimester of pregnancy, while the control group received routine breastfeeding education as part of standard antenatal care. Data were collected before and after the educational intervention.

The primary focus of the study was to compare changes in breastfeeding self-efficacy and infant feeding attitudes between the two groups following the intervention. The findings of this study are expected to contribute to the growing evidence on the use of innovative digital and gamification-based educational approaches in antenatal breastfeeding education.

DETAILED DESCRIPTION:
This randomized controlled study was designed to evaluate the effectiveness of a gamification-based digital breastfeeding education program on breastfeeding self-efficacy and infant feeding attitudes among pregnant women. The study was conducted at the Obstetrics and Gynecology outpatient clinics of Lokman Hekim Etlik Hospital, where pregnant women are routinely followed during the antenatal period.

After being informed about the purpose and procedures of the study, pregnant women who agreed to participate provided written and verbal informed consent. Participants were allocated to the intervention or control group using a block randomization method to ensure balanced group sizes. The randomization sequence was generated by an independent statistician, and group assignments were concealed using sequentially numbered, opaque sealed envelopes. This process was implemented to reduce selection bias and strengthen the internal validity of the study.

The intervention consisted of a structured breastfeeding education program delivered through a digital platform incorporating gamification elements. The educational content was designed to increase participant engagement and motivation by integrating interactive and game-based components into standard breastfeeding education. The program was administered during the last trimester of pregnancy and focused on enhancing confidence in breastfeeding and fostering positive infant feeding attitudes.

Participants in the control group received routine breastfeeding education provided as part of standard antenatal care services at the hospital. This education reflected usual clinical practice and did not include digital or gamification-based components.

Data collection was conducted at baseline and following completion of the educational intervention. The study evaluated changes in breastfeeding-related psychosocial outcomes by comparing pre- and post-intervention assessments between the intervention and control groups.

This study aims to contribute to the evidence base on innovative digital education strategies in maternal health by examining the potential benefits of gamification-enhanced breastfeeding education during pregnancy. The findings are expected to support the development of engaging, technology-supported antenatal education programs to improve breastfeeding preparedness.

ELIGIBILITY:
Inclusion Criteria:

* Primipara,
* Between 27-40 weeks of gestation,
* Those who have not received breastfeeding training before,
* Able to speak and understand Turkish,
* Women with a smart phone/tablet/computer with internet connection will be included in the study.

Exclusion Criteria:

* Having a high risk pregnancy
* with a condition that prevents breastfeeding
* fetus with abnormality

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2023-03-30 (Actual); Study Completion 2023-05-30 (Actual)

PRIMARY OUTCOMES:
breastfeeding self-efficacy | One week before the intervention and two weeks after completion of the intervention.
  Breastfeeding self-efficacy was measured using the Breastfeeding Self-Efficacy Scale-Short Form, Antenatal Version (BSES-SF). The scale consists of 14 items with total scores ranging from 14 to 70. Higher scores indicate greater breastfeeding self-efficacy.
infant feeding attitudes | One week before the intervention and two weeks after completion of the intervention.
  Infant feeding attitudes were assessed using the Iowa Infant Feeding Attitude Scale (IIFAS). The scale includes 17 items with total scores ranging from 17 to 85. Higher scores reflect more positive attitudes toward breastfeeding.

CONTACTS AND LOCATIONS:
Locations (1):
- Lokman Hekim University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
This study will be conducted to determine the effect of breastfeeding education given through gamification on breastfeeding self-efficacy and infant feeding attitudes of pregnant women.